CLINICAL TRIAL: NCT00468910
Title: Spectral Markers in Aspirin Chemoprevention of Colonic Neoplasia
Brief Title: Aspirin in Preventing Colorectal Cancer in Patients at Increased Risk of Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00841; NCI-2009-00841 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000652929; NCI 04-2-03 (Other: Northwestern University); NWU04-2-03 (Other: DCP); N01CN35157 (NIH)
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Colon Cancer; Precancerous Condition; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Precancerous Conditions; Rectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral acetylsalicylic acid (aspirin) once daily.
  Interventions: Drug: acetylsalicylic acid; Other: laboratory biomarker analysis
- Arm II (Placebo Comparator): Patients receive oral placebo once daily.
  Interventions: Drug: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: acetylsalicylic acid — Given orally
  Other Names: ASA; Ecotrin; Empirin; Extren
  Arms: Arm I
Drug: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II
Other: laboratory biomarker analysis — Correlative study

SUMMARY:
This randomized phase II trial is studying how well aspirin works in preventing colorectal cancer in patients at increased risk of colorectal cancer. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of aspirin may prevent colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine whether acetylsalicylic acid (aspirin) will alter spectral markers (i.e., spectral slope and fractal dimension) in distal colonic mucosa of patients who are at increased risk for the development or recurrence of colorectal cancer.

SECONDARY OBJECTIVES:

I. Assess the effect of this drug on colonic epithelial apoptosis and cell proliferation in these patients.

II. Assess the effect of this drug on rectal prostaglandin levels in these patients.

III. Assess the effect of this drug on platelet cyclooxygenase activity in these patients.

IV. Correlate changes in spectral markers with UGT1A6 genotype in patients treated with this drug.

OUTLINE: This is a multicenter, randomized, double-blind, placebo-controlled study. Patients are stratified by clinical site and adenoma/carcinoma maximal size. Patients with abnormal spectral biomarkers are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral acetylsalicylic acid (aspirin) once daily.

ARM II: Patients receive oral placebo once daily.

In both arms, treatment continues for 3 months in the absence of unacceptable toxicity.

Patients undergo flexible sigmoidoscopy and biopsies as well as blood collection at baseline (during prestudy colonoscopy) and at completion of study treatment for comparison of spectral signatures with biomarkers of both aspirin activity (including plasma cyclooxygenase activity and rectal prostaglandin levels) as well as with biomarkers associated with antineoplastic alteration (including apoptosis and cell proliferation). UGT1A6 genotyping analysis is also performed.

After completion of study treatment, patients are followed at 3 months.

ELIGIBILITY:
Criteria:

* No active or metastatic cancer within the past 6 months
* Scheduled to undergo colonoscopy for colonic neoplasia surveillance
* Hemoglobin >= 12.0 g/dL
* Platelet count >= 120,000/mm^3
* AST or ALT =< 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase =< 1.5 times ULN
* Bilirubin =< 1.5 times ULN
* BUN =< 40 mg/dL
* Glomerular filtration rate >= 45 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No coagulopathy
* No anemia
* No history of peptic ulcer disease or gastrointestinal hemorrhage
* No history of cerebrovascular accident
* No uncontrolled hypertension
* No history of intolerance or allergy to aspirin or to NSAIDs
* No liver disease as manifested by signs or symptoms of cirrhosis
* No endoscopic or radiographic evidence of portal hypertension
* No active colitis by endoscopy
* No history of inflammatory bowel disease
* No requirement for aspirin as medical therapy (i.e., post-myocardial infarction or transient ischemic attack)
* No untreated helicobacter pylori infection
* History of significant colonic neoplasia, defined as 1 of the following:

  * Adenoma within the past 6 years
  * Colorectal cancer within the past 6 years
  * Known adenoma on present exam
  * Histologically confirmed polyps seen on imaging
* INR =< 1.5
* At least 6 months since prior cancer treatment
* No other concurrent acetylsalicylic acid (aspirin)-containing products or non-steroidal anti-inflammatory drugs (NSAIDs)
* No concurrent systemic corticosteroids
* No other concurrent anticoagulants or antiplatelet agents
* No concurrent investigational drugs

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hemant Roy, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Roy HK, Turzhitsky V, Wali R, Radosevich AJ, Jovanovic B, Della'Zanna G, Umar A, Rubin DT, Goldberg MJ, Bianchi L, De La Cruz M, Bogojevic A, Helenowski IB, Rodriguez L, Chatterton R, Skripkauskas S, Page K, Weber CR, Huang X, Richmond E, Bergan RC, Backman V. Spectral biomarkers for chemoprevention of colonic neoplasia: a placebo-controlled double-blinded trial with aspirin. Gut. 2017 Feb;66(2):285-292. doi: 10.1136/gutjnl-2015-309996. Epub 2015 Oct 26. PMID 26503631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual 02/22/2007 and closed to accrual 08/10/2009. Subjects were recruited at Northwestern University and University of Chicago.
Pre-assignment Details: A total of 110 subjects met the clinical definition of high risk for colorectal cancer, were entered onto the trial, and underwent initial spectral analysis. Of these, 81 had a cancer-associated spectral signature in histologically normal colonic mucosa.79 of these 81 subjects were randomized and began the study intervention
Groups:
- Acetylsalicylic Acid: Patients receive oral acetylsalicylic acid (aspirin) once daily.
- Placebo: Patients receive oral placebo once daily.
Period: Overall Study
Arm/Group | Acetylsalicylic Acid | Placebo
Started | 40 | 39
Randomization | 40 | 39
Treatment | 36 | 36
Post-Treatment Biopsy | 36 | 36
Follow-up | 36 | 36
Completed | 36 | 36
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Medical Contraindication | 0 | 1

BASELINE CHARACTERISTICS:
Population: 72 of the 79 subjects who were randomized completed the primary endpoint (3-month tissue biopsy); 36 from each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetylsalicylic Acid | Placebo | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 34 | 67
  >=65 years | 7 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 25 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 37 | 39 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 37 | 36 | 73
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of a Spectral Biomarker for Colonic Carcinogenesis (Called Spectral Slope or SPEC) From Baseline to 3 Months.
Description: Spectral marker assessment was performed via LEBS analysis (low-coherence enhanced backscattering spectroscopy) on the uninvolved mucosal biopsies of subjects taken at baseline and after 3 months of treatment with either aspirin or placebo. SPEC characterizes the size distribution of macromolecular complexes and other intracellular structures, with a decrease of the spectral slope implying a shift of the size distribution of intracellular structures toward smaller sizes.
  Spectral markers SPEC and FRAC provide a measure of the fundamental characteristics of the tissue nanoscale architecture.
Time Frame: 3 months from baseline colonoscopy to end of intervention.
Population: Subjects at high risk for colorectal cancer (CRC) with a cancer-associated spectral marker signature in histologically normal colonic mucosa.
Measure: Mean (Standard Deviation); unit: micron^-1
Groups:
- Acetylsalicylic Acid: Patients receive oral acetylsalicylic acid (aspirin) 325 mg once daily.
Arm/Group | Acetylsalicylic Acid | Placebo
Number analyzed (Participants) | 36 | 36
micron^-1
  Baseline | 40.72 (16.91) | 37.54 (21.64)
  Post Intervention | 43.45 (26.84) | 37.52 (28.15)
Statistical Analysis 1: Comparison: Acetylsalicylic Acid vs Placebo; The study was powered to detect an attributable change in the aspirin group of 50% relative to baseline values - an approximate 50% increase in spectral slope; Test type: Superiority or Other; p = 0.11, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change of a Spectral Biomarker for Colonic Carcinogenesis (Called Fractal Dimension or FRAC) From Baseline to 3 Months.
Description: Spectral marker assessment was performed via LEBS analysis (low-coherence enhanced backscattering spectroscopy) on the uninvolved mucosal biopsies of subjects taken at baseline and after 3 months of treatment with either aspirin or placebo. FRAC characterizes the spatial autocorrelation function of mass density distribution in tissue.
  SPEC and FRAC provide a measure of the fundamental characteristics of the tissue nanoscale architecture
Time Frame: 3 months from baseline colonoscopy to end of intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Acetylsalicylic Acid | Placebo
Number analyzed (Participants) | 36 | 36
unitless
  Baseline | 142.41 (2570.86) | 23.28 (2699.82)
  Post Intervention | -407.78 (3470.69) | 650.97 (3201.77)
Statistical Analysis 1: Comparison: Acetylsalicylic Acid vs Placebo; Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Colonic Epithelial Apoptosis as Measured by Immunohistochemical Detection of Cleaved Caspase 3
Description: Evaluate the effect of aspirin on colonic epithelial apoptosis and cell proliferation as assessed by immunohistochemical detection of cleaved caspase 3 .These were performed on samples that had been previously analyzed for 4D-ELF.
Time Frame: 3 months from baseline colonoscopy to end of intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Total Cells
Arm/Group | Acetylsalicylic Acid | Placebo
Number analyzed (Participants) | 36 | 36
Percentage of Total Cells
  Baseline | 4.56 (4.27) | 5.24 (3.69)
  At 3 Months | 4.26 (4.44) | 7.26 (6.77)

4. Secondary Outcome: Changes in Colonic Cell Proliferation as Measured by Immunohistochemical Detection of Ki67
Description: Evaluate the effect of aspirin on colonic epithelial apoptosis and cell proliferation as assessed by immunohistochemical detection of Ki-67. These were performed on samples that had been previously analyzed for 4D-ELF.
Time Frame: 3 months from baseline colonoscopy to end of intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Total Cells
Arm/Group | Acetylsalicylic Acid | Placebo
Number analyzed (Participants) | 36 | 36
Percentage of Total Cells
  Baseline | 38.07 (16.83) | 40.45 (12.26)
  3 Months Intervention | 43.60 (14.77) | 37.74 (13.37)

5. Secondary Outcome: Rectal Prostaglandin Levels as Measured by ELISA
Description: Evaluate the effect of aspirin on rectal prostaglandin levels.
Time Frame: 3 months from baseline colonoscopy to end of intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Acetylsalicylic Acid | Placebo
Number analyzed (Participants) | 36 | 36
pg/ml
  Baseline | 305.93 (300.01) | 654.64 (1536.52)
  Post Intervention | 211.97 (134.32) | 209.02 (134.33)

6. Other Pre Specified Outcome: Platelet Cyclooxygenase (COX) Activity as Measured by a Peroxidase-based COX Enzyme Activity Assay
Description: Evaluate the effect of aspirin on platelet COX activity as measured by a peroxidase-based Cox enzyme activity assay.
Time Frame: 3 months from baseline colonoscopy to end of intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Acetylsalicylic Acid | Placebo
Number analyzed (Participants) | 36 | 36
pg/ml
  Baseline | 712976.73 (2082413.36) | 430109.56 (798782.31)
  Post Intervention | 6914.87 (20891.41) | 200233.5 (463029.1)

ADVERSE EVENTS:
Time Frame: 3 months from baseline colonoscopy to end of intervention and repeat colonoscopy.
Groups:
- Acetylsalicylic Acid: Patients receive oral acetylsalicylic acid (aspirin) once daily.
  acetylsalicylic acid: Given orally
  laboratory biomarker analysis: Correlative study
- Placebo: Patients receive oral placebo once daily.
  placebo: Given orally
  laboratory biomarker analysis: Correlative study
Arm/Group | Acetylsalicylic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 17/40 | 21/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetylsalicylic Acid (N=40) | Placebo (N=39)
Blood/Bone Marrow: Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (3)
Blood/Bone Marrow: Other (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Hemorrhage with Surgery (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain: Stomach (General disorders) | 2 (2) | 2 (2)
Pain: Abdomen Nos (General disorders) | 2 (2) | 1 (2)
Pain: Head/Headache (General disorders) | 1 (1) | 4 (4)
Pain: Other (General disorders) | 1 (1) | 1 (1)
Pain: Joint (General disorders) | 0 (0) | 1 (1)
Pain: Extremity - Limb (General disorders) | 0 (0) | 1 (1)
Pain: Uterus (General disorders) | 0 (0) | 1 (1)
Constitutional Symptoms: Fever (General disorders) | 0 (0) | 1 (1)
Constitutional Symptoms: Insomnia (General disorders) | 0 (0) | 1 (1)
Constitutional Symptoms: Weight Gain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constitutional Symptoms: Other (General disorders) | 0 (0) | 1 (1)
Rhinitis (Immune system disorders) | 1 (1) | 0 (0)
Upper Airway Nos (Infections and infestations) | 1 (1) | 2 (2)
Infection - Other (Infections and infestations) | 0 (0) | 2 (2)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
AST (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ALT (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (2)
Sexual - Other (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less